CLINICAL TRIAL: NCT01465269
Title: Treatment of Social Competence in Military Veterans, Service Members, and Civilians With Traumatic Brain Injury
Brief Title: Treatment of Social Competence After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: Rehabilitation Hospital of Indiana (Other); Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); Wayne State University (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Cynthia Harrison-Felix, PhD, Assistant Director of Research, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT100068
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Social Competence
MeSH Terms: conditions — Brain Injuries, Traumatic; Social Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GIST Intervention (Experimental)
  Interventions: Behavioral: Group Interactive Structured Treatment
- Alternative Intervention (Active Comparator)
  Interventions: Behavioral: Alternative Intervention

INTERVENTIONS:
Behavioral: Group Interactive Structured Treatment — GIST groups consist of 8 group participants and two group therapists. Group members receive the workbook and are asked to bring it to each session. During each of the 13, 1.5 hour sessions, key concepts from the previous session are reviewed, a new topic is discussed, strategies and skills are practiced interactively, and real-life social problems are addressed. Previously covered topics are integrated into each session through discussion and problem solving to provide repetition and reinforcement of information.
  Arms: GIST Intervention
Behavioral: Alternative Intervention — Participants in the alternative treatment will attend 13 weekly classroom sessions, where they will view video presentations of the same curriculum topics covered in the GIST workbook. The group therapists will serve as moderators and will meet with participants individually. Group interaction will not be encouraged. Homework exercises will be offered but participants will not be asked to return their homework and will not receive any feedback.
  Arms: Alternative Intervention

SUMMARY:
The aim of this study is to determine the effectiveness of holistic group treatment program (called Group Interactive Structured Treatment, or GIST) to improve social communication skills for individuals with Traumatic Brain Injury. Hypothesis: Compared to an alternative intervention, those receiving the GIST intervention will show improved social competence, improved quality of life, and stronger group cohesion.

DETAILED DESCRIPTION:
Background: Impairments in social competence are among the most prevalent sequelae after traumatic brain injury (TBI). Without successful social skills a person is often isolated, in conflict with others, and denied access to social and vocational opportunities. The aim of this study is to determine the effectiveness of a manualized group treatment program to improve and maintain social competence for individuals with TBI with identified social skill deficits. The Group Interactive Structured Treatment (GIST) - Social Competence program is a holistic, dual-disciplinary intervention targeting the pervasive interpersonal and communication problems that often interfere with participation at work, home, school and in the community after TBI.

Aims and Hypotheses: Aim 1: Measure the effectiveness of the GIST intervention with multisite implementation. Hypothesis 1a: Those receiving the GIST will demonstrate significant improvement in social competence, compared to those receiving the alternative treatment, as measured by the Profile of Pragmatic Impairment in Communication (PPIC). Hypothesis 1b: Compared to the alternative intervention, those receiving the GIST will maintain improvement in social competence at 3 months post-intervention, as measured by the PPIC. Hypothesis 1c: Compared to the alternative intervention, those receiving the GIST will demonstrate improvement in additional aspects related to social competence at 3 months post-intervention, as measured by the LaTrobe Communication Questionnaire, the Goal Attainment Scale, the Brief Symptom Inventory-18, and the Post Traumatic Stress Disorder Check List - Civilian version. Hypothesis 1d: Compared to the alternative intervention, those receiving the GIST will demonstrate improvement at 3 months post intervention in quality of life, as measured by the Satisfaction with Life Scale. Aim 2: Identify the potent ingredients associated with the GIST. Hypothesis 2a: FOr participants in the GIST intervention, higher group cohesion measured by the TFI: Cohesiveness Scale will be associated with improved social competence. Hypothesis 2b: Compared to the alternative intervention, those receiving the GIST will demonstrate stronger social self efficacy associated with improved social competence, as measured by the Scale of Perceived Self Efficacy.

Study Design: This study uses a two-arm, multi-centered randomized controlled clinical trial design to compare the GIST treatment to an alternative treatment, in which participants are presented information from the GIST treatment program without the group process. A total of 192 military, veteran and civilian participants with mild to moderate TBI will be enrolled by six centers. Measures will be collected at baseline, post-treatment, and 3 months post-treatment. Videotapes of participants will be evaluated for social competence by blinded independent raters, and progress on individualized social skills goals will be assessed. Replicable training of group leaders will include a 2 ½ day in-person workshop followed by feedback during a pilot of the intervention and alternative intervention. The fidelity of the intervention will be assessed by independent raters using a standardized instrument to ensure that the intervention is implemented consistently. Results of this study will be disseminated to relevant stakeholders via presentations and publications. By the end of this study, the field will have definitive evidence about the effectiveness of a group social competence intervention for people with TBI.

Military Benefit: The proposed study has a high degree of relevance for returning OIF/OEF soldiers and veterans post-TBI due to the prevalence of social reintegration difficulties in this population. The GIST intervention has the potential to assist our soldiers and veterans in returning to full participation in their families, communities and productive activity.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of a TBI as evidenced by self report on OSU TBI ID screen
* Sustained a TBI anytime after October 2001;
* are at least 6 months post injury
* score at Level 1 (Independent) or Level 2 (Overnight Supervision) on the Supervision Rating Scale;
* are 18 years of age or older at the time of the study;
* have adequate receptive/expressive communication skills functional for group participation, (score >5 on the Comprehension and Expression of the Functional Independence Measure (FIM)70 based on results of screening interview;
* possess the English language skills necessary to participate in the group intervention and complete study measures;
* demonstrate some aspect of problematic social competence by responding "yes" to at least one of 5 screening statements listed here, as reported by the participant or their support person.
* provide Informed Consent to participate.

Exclusion Criteria:

* are unable to verbally communicate, or require augmentative communication system;
* are unable to attend the majority of group sessions (e.g., living at a distance from the site without consistent transportation; going on an extended vacation, planned surgeries, planning to move);
* are currently involved in ongoing structured group psycho-social therapy;
* are currently participating in another clinical trial.
* are currently in one-on-one therapy with one of the therapists
* have already participated in the GIST intervention
* in the opinion of the PI, have any conditions which might interfere with complete of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Profile of Pragmatic Impairment in Communication (PPIC) | Baseline, 13 weeks (post-treatment), 25 weeks (3 mos post-treatment)
  This tool is designed to measure social communication impairments following TBI. It focuses not only on communication skills but also on other aspects of socially competent behavior, such as social perception and adherence to social boundaries. Videotaped conversations at the 3 time points will be evaluated using the PPIC to assess change from baseline.

SECONDARY OUTCOMES:
Change from Baseline on LaTrobe Communication Questionnaire (LCQ) | Baseline, 13 weeks (post-treatment), 25 weeks (3-mos post-treatment)
  A 30-item questionnaire that measures cognitive-communication ability, a subjective secondary outcome measure.
Change from baseline on Goal Attainment Scale | 3 weeks into intervention, 13 weeks (post-intervention), 25 weeks (3-mos post-intervention)
  A flexible system of measuring outcome goals in individuals with TBI, based on a five-point scale. Levels of goal attainment are expressed objectively in terms of concrete behaviors that can be observed and recorded
Change from Baseline on Brief Symptom Inventory-18 | Baseline, 13 weeks (post treatment), 25 weeks (3 mos post-treatment)
  Consists of 18 emotional distress items that are rated on a 5 point Likert scale and yields a Global Severity Index as well as Somatic, Anxiety, and Depressive Dimension scores.
Change from Baseline on Satisfaction with Life Scale | Baseline, 13 weeks (post-treatment), 25 weeks (3 mos post-treatment)
  A subjective, 5-item scale of self-rating of global life satisfaction

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Polytrauma Rehabilitation Center, Palo Alto, California
  - Craig Hospital, Englewood, Colorado
  - Rehabilitation Hospital of Indiana, Indianapolis, Indiana
  - Rehabilitation Institute of Michigan, Detroit, Michigan
  - Hunter Holmes McGuire Medical Center, Richmond, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Harrison-Felix C, Newman JK, Hawley L, Morey C, Ketchum JM, Walker WC, Bell KR, Millis SR, Braden C, Malec J, Hammond FM, Eagye CB, Howe L. Social Competence Treatment After Traumatic Brain Injury: A Multicenter, Randomized Controlled Trial of Interactive Group Treatment Versus Noninteractive Treatment. Arch Phys Med Rehabil. 2018 Nov;99(11):2131-2142. doi: 10.1016/j.apmr.2018.05.030. Epub 2018 Jun 30. PMID 29966645